CLINICAL TRIAL: NCT02319434
Title: Validating the Use of a Novel Wearable Device in Improving Quality of Life of Ostomy Patients
Brief Title: Ostom-i Alert Sensor Quality of Life Validation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Associate Professor, Department of Anesthesiology, Pain, and Perioperative Medicine, Stanford University
Other Study IDs: IRB-32211
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Ostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ostom-i Alert Sensor — Sensor on ostomy bag.

SUMMARY:
The purpose of this study is to determine the usability and acceptance of the Ostom-i Alert Sensor. The investigators would like to see if is generally helpful to ostomy patients and whether it has a beneficial impact on living with an ostomy bag. Results from this study will be used to determine if a larger clinical study is feasible.

DETAILED DESCRIPTION:
Evidence from clinical experience shows that patients with ostomies go through a significant life change to learn to live with the ostomy bag. These changes can include "an altered body image, changes in daily routines, and for some, changes in life patterns such as work and leisure activities" (Burckhardt). Previous studies have also shown that ostomy patients have negative changes in their physical, psychological, social, and spiritual quality of life (Krouse).

An ostomy patient developed the Ostom-i Alert Sensor after experiencing these changes - the goal of the sensor is to make life easier for patients with ostomy bags, by allowing for easier output measurements and anticipation of bag changes. In this study, we hope to use this new device and track any improvements for quality of life for ostomy patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* use of an ostomy bag for at least six months
* must own an iPhone, iPod Touch, or Android

Exclusion Criteria:

* use of large urostomy bags

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be seeking participants from communities of ostomy patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Improved quality of life with any ostomy bag | 4 weeks
  We would like to see if using the sensor improves the quality of life while living with an ostomy bag.

SECONDARY OUTCOMES:
Self-management (able to manage using and changing their ostomy bag) | 4 weeks
  Are users better able to manage using and changing their ostomy bag?
Sleep quality (report a higher quality of sleep while using the sensor with their ostomy bag?) | 4 weeks
  Do participants report a higher quality of sleep while using the sensor with their ostomy bag?
Confidence and self-image (participant report a better self-image and more self-confidence?) | 4 weeks
  Do participants report a better self-image and more self-confidence with their ostomy bag than before using the sensor?

CONTACTS AND LOCATIONS:
Overall Officials: Larry F Chu, MD, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burckhardt CS. The Ostomy Adjustment Scale: Further evidence of reliability and validity. Rehabilitation Psychology 35(3): 149-155, 1990.
- [Background] Krouse R, Grant M, Ferrell B, Dean G, Nelson R, Chu D. Quality of life outcomes in 599 cancer and non-cancer patients with colostomies. J Surg Res. 2007 Mar;138(1):79-87. doi: 10.1016/j.jss.2006.04.033. Epub 2006 Dec 29. PMID 17196990
- [Background] Grant M, Ferrell B, Dean G, Uman G, Chu D, Krouse R. Revision and psychometric testing of the City of Hope Quality of Life-Ostomy Questionnaire. Qual Life Res. 2004 Oct;13(8):1445-57. doi: 10.1023/B:QURE.0000040784.65830.9f. PMID 15503840
- [Derived] Rouholiman D, Gamble JG, Dobrota SD, Encisco EM, Shah AG, Grajales Iii FJ, Chu LF. Improving Health-Related Quality of Life of Patients With an Ostomy Using a Novel Digital Wearable Device: Protocol for a Pilot Study. JMIR Res Protoc. 2018 Mar 26;7(3):e82. doi: 10.2196/resprot.7470. PMID 29581087